CLINICAL TRIAL: NCT02189291
Title: When to Remove the Indwelling Catheter After Minimally Invasive Sacrocolpopexy?
Brief Title: Study to Assess Duration of Indwelling Catheter After Sacrocolpopexy
Acronym: CARESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, W. Thomas Gregory, Associate Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 00010603
Record Dates: First submitted 2014-07-03; First posted 2014-07-14 (Estimated); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Pelvic Organ Prolapse; Urinary Tract Infections; Urinary Retention
Keywords: Indwelling catheter; Hospital stay; Urinary tract infection; Sacrocolpopexy
MeSH Terms: conditions — Pelvic Organ Prolapse; Urinary Tract Infections; Urinary Retention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate catheter removal (Experimental): The indwelling Foley catheter will be removed prior to exiting the operating room.
  Interventions: Procedure: Immediate catheter removal
- Post op day 1 catheter removal (Active Comparator): Patients assigned to this group will follow the standard of care at present, with removal of indwelling catheter on the morning of postoperative day 1.
  Interventions: Procedure: Post op day 1 catheter removal

INTERVENTIONS:
Procedure: Immediate catheter removal — The indwelling catheter will be removed prior to exiting the operating room.
  Arms: Immediate catheter removal
Procedure: Post op day 1 catheter removal — For patients assigned to catheter removal on post operative day one, which is the standard of care at this point.
  Arms: Post op day 1 catheter removal

SUMMARY:
Objectives

The objective of this study is to help identify the best practice regarding the use of indwelling catheter after minimally invasive urogynecologic surgery. Investigators propose a randomized controlled trial comparing the immediate removal of indwelling urethral catheter, after minimally invasive sacrocolpopexy, to the present standard catheter removal on post operative day one. Evidence based catheter management will be helpful to both providers and patients in post-operative decision making.

Specific Aims

Aim 1: To demonstrate that immediate removal of catheter after minimally invasive sacrocolpopexy results in shorter hospital stay than removal on postoperative day 1.

Aim 2: To demonstrate that immediate removal of catheter after minimally invasive sacrocolpopexy confers no increased risk of re-catheterization.

Aim 3: To demonstrate that immediate removal of catheter after minimally invasive sacrocolpopexy decreases the occurrence of urinary tract infection.

Design

A randomized controlled trial comparing the standard overnight indwelling urethral catheterization with removal of catheter immediately post surgery after minimally invasive sacrocolpopexy, at Oregon Health & Science University.

Outcome measures

Primary outcome measures are hospital stay in hours after completion of surgery and need for re-catheterization. Hospital stay will be counted from the time the patient leaves the operating room to the time she leaves the hospital. To avoid confounding, investigators are only including the first / morning case of the day. For re-catheterization, investigators will evaluate if patient was able to void after completion of surgery. Investigators will compare the post voiding residuals, the need for re-catheterizations and the numbers of patients going home with an indwelling catheter between the two groups. Investigators will also compare the number of urinary tract infections, as documented by urine culture and subsequent treatment, between the two groups.

Study Subjects

Study subjects will be women undergoing minimally invasive sacrocolpopexy. Women will be invited to participate in the study during their preoperative visit. If they agree to participation, this will be noted in their chart. Randomization to group will occur immediately following surgery.

DETAILED DESCRIPTION:
Objectives

The objective of this study is to help identify the best practice regarding the use of indwelling catheter after minimally invasive urogynecologic surgery. Investigators propose a randomized controlled trial comparing the immediate removal of indwelling urethral catheter, after minimally invasive sacrocolpopexy, to the present standard catheter removal on post operative day one. Evidence based catheter management will be helpful to both providers and patients in post-operative decision making.

Specific Aims

Placement of indwelling catheter after minimally invasive pelvic organ prolapse (POP) surgery is routine practice. There is limited evidence to support the use of overnight indwelling catheters, and despite this, the use of catheters after urogynecologic surgery remains common practice. The objective of this study is to help identify the best practice regarding the use of indwelling catheter after minimally invasive urogynecologic surgery. Dunn et al found that immediate removal of catheter after completion of an uncomplicated abdominal or vaginal hysterectomy was not associated with re-catheterization, urinary tract infections or fever. They also found that patients in whom the catheter was removed immediately had less pain compared to the patients who had indwelling catheter for 24 hours. The applicability of this study to Urogynecology is limited by the fact that patients with incontinence and / or prolapse were not included in it. Use of catheters after surgery may be convenient for providers, but the benefit to the patient is uncertain. Investigators believe that evidence with regards to the optimal use of catheter use in urogynecologic surgery will be helpful to the providers.

Risk of urinary tract infection increases the longer an indwelling catheter stays in a patient. Urinary tract infections associated with catheters (CAUTI) are responsible for 40% of hospital acquired infections. CAUTI are associated with 387, 550 hospital acquired infections in a year, which could be prevented. Investigators believe that avoiding placement of catheter after minimally invasive urogynecologic surgery will result in shorter hospital stay and reduction in CAUTI, thereby improving the quality and cost of health care.

Aim 1: To demonstrate that immediate removal of catheter after minimally invasive sacrocolpopexy results in shorter hospital stay than removal on postoperative day 1.

Aim 2: To demonstrate that immediate removal of catheter after minimally invasive sacrocolpopexy confers no increased risk of re-catheterization.

Aim 3: To demonstrate that immediate removal of catheter after minimally invasive sacrocolpopexy decreases the occurrence of urinary tract infection.

Background

Most patients stay in hospital for a 23-hour observation following minimally invasive urogynecologic surgery. The usual practice is to leave the indwelling urethral catheter overnight after these procedures. The use of indwelling catheters after surgery is carried for multiple reasons, including measuring urinary output and prevention of urinary retention after surgery. The use of indwelling Foley catheter after surgery is associated with prolonged hospital stay, fever and urinary tract infection. A study by Haakvort et al compared removal of indwelling catheter on post operative day 1 to longer catheterization after vaginal and found a tenfold reduction in urinary tract infections.

The removal of indwelling catheter may affect the length of stay in hospital, with associated budgetary and economic implications. One study found that removal of indwelling catheter at midnight results in patients being discharged 0.7 days earlier than patients who had their catheters removed in the morning. This results in shorter length of hospital stay and improved discharge planning. There is a wide variation in practice and policies regarding catheter removal. With no clear evidence-based practice regarding catheter removal, and lack of data in literature with regards to catheter removal after urogynecologic surgery, practices vary among physicians and institutions. Audits in British hospitals found that almost half of the catheters were removed either at the discretion of the nurse or at the time of rounds in the morning. Another study found that when the catheters were scheduled to be removed in the morning, only 70% were removed in time.

Dunn et al looked into removal of indwelling catheter immediately after hysterectomy compared to removal after 24 hours. They found that immediate removal of catheter after surgery was not associated with any adverse outcomes or need for re-catheterization, and patients with immediate removal reported significantly less pain compared to their counterparts who had catheter removal at 24 hours. Similarly, Alessandri found that women who had their catheter removed early had a shorter mean ambulation time and their hospital stay was shorter by 19 hours. This shows the economic benefit with early discharge associated with early catheter removal, however such a study is lacking in urogynecology literature.

In addition to potential benefits to health care costs, immediate catheter removal has several health benefits. There is evidence that early ambulation reduces the incidence of clinically evident deep venous thrombosis. Therefore, early removal of indwelling urethral catheter after surgery may contribute towards reducing postoperative morbidity by reducing the incidence of post operative deep venous thrombosis and decrease health care cost by aiding towards early discharge. Another advantage of immediate catheter removal after surgery is lower incidence of urinary tract infection.

There are few studies offering insight into postoperative voiding efficiency after uncomplicated minimally invasive urogynecologic surgery. There is variation in practice with regards to the length of time the indwelling catheter is left in place. Multiple factors contribute to how long a catheter stays. In the absence of strong evidence, this decision depends on physician preference, staff convenience and patient tolerance. The use of indwelling urethral catheter is the usual practice after gynecologic and POP surgery. Despite this routine practice, there seems to be little evidence supporting the use of indwelling urethral catheter after gynecologic surgery. Generally, the indwelling urethral catheter is used after surgery for monitoring output, or if the patient is not mobile. This may not be the usual case after urogynecologic surgery. Some of the reasons for routine use of catheter after urogynecologic surgery include allowing bladder emptying as voiding may be difficult due to the effects of the surgery, such as pain or swelling of surrounding soft tissues. The routine use of indwelling catheters after routine urogynecologic surgery carries the risk of morbidity including detrusor overactivity, urinary tract infection or pain in urethra.

There is a lack of agreement among providers regarding the optimal time for removal of urethral catheter after surgery. Usual practices are based on provider preference and the already established institution practices rather than evidence based practice. Although different institutions and providers have different practices and policies, there is no evidence based practice regarding the effect of the time when catheter is removed or for the length of time catheter is left in place prior to removal after surgery. Most places will leave the catheter overnight after surgery. One possible reason for that may be that the reduced staff at night may not respond to the complication of urinary retention, following catheter removal. Another perceived reason for leaving the catheter in overnight is that patients will rest through the night and then get back to their normal voiding the next day, once the catheter is removed in the morning. Cochrane review by Griffiths and Fernandez had suggested the need for randomized trials to address questions regarding catheter removal among discrete subgroups and specialties. The usual practice of indwelling foley catheter after urogynecologic surgery may be convenience to the providers, but there is limited evidence in literature regarding what benefits patients gain from this practice.

Outcome measures

Primary outcome measures are hospital stay in hours after completion of surgery and need for re-catheterization. Hospital stay will be counted from the time the patient leaves the operating room to the time she leaves the hospital. To avoid confounding, investigators are only including the first / morning case of the day. For re-catheterization, investigators will evaluate if patient was able to void after completion of surgery. Investigators will compare the post voiding residuals, the need for re-catheterizations and the numbers of patients going home with an indwelling catheter between the two groups. Investigators will also compare the number of urinary tract infections, as documented by urine culture and subsequent treatment, between the two groups.

Data Collection

Investigators will obtain demographic information. On post operative day 1, investigators will obtain patient satisfaction and pain scores. Pain score will be obtained with the use of pictorial "Wong Scale," assessing level of pain and location (i.e., bladder or urethra vs. the surgical site). Furthermore, patients will be asked whether they will use the same treatment again (yes or no).

All patients are to expect discharge the following day and counseled as such. Patients assigned to immediate removal will undergo the following protocol: The indwelling catheter will be removed prior to exiting the operating room. If the patient has an urge to void immediately post operatively, the void will be recorded and post void residual determined by bladder scan. If the post void residual is no more than 1/3 of the total volume, the patient will be considered to have passed the voiding trial and have no further intervention. In patients with more than 1/3 post void residual or inability to void four hours after completion of surgery, bladder volume will be checked with a bladder scan. In subjects with less than 300 mL of urine, they will be given an additional two hours to void. For patients with >300 mL of urine, they will undergo straight catheterization and re-enter the voiding trial cycle. For patients who have not voided at six hours, straight catheterization will be performed and they will re-enter the voiding trial cycle and given four hours to void. This process will continue for three total cycles (1st cycle post operative, two cycles thereafter), at which time they will be given an indwelling catheter.

For patients assigned to catheter removal on post operative day one, investigators will perform backfill voiding trial prior to catheter removal. Investigators are planning to perform backfill voiding trial as it has not been shown to be inferior to waiting to void and this will avoid confounding regarding the discharge time from hospital. Bladder will be filled with 300 mL of sterile water and the indwelling catheter will then be removed. Patient will be asked to void in a hat thereafter, if they are able to void at least 200 mL, they would have completed a successful voiding trial. If they are unable to void, then investigators will perform straight catheterization and allow them four hours to void. Patients unable to pass the voiding trial after two attempts will go home with either an indwelling catheter or performing self catheterization (depending on patient's comfort). For the purpose of the study, patients going home with a catheter or self catheterization will be in the same group of going home with a catheter. Investigators will compare the incidence of urinary tract infections within four weeks after surgery, as documented by urine culture and / or treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing minimally invasive sacrocolpopexy
* Sacrocolpopexy with or without concomitant procedures
* Patients having the first start surgery of the day to standardize hospital time.

Exclusion Criteria:

* Elevated post void residual (PVR)
* Mobility problems
* Neurological conditions
* Intra-operative cystotomy or urinary tract injury

Ages: 21 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Hospital stay | 4 weeks
  Primary outcome measure is hospital stay in hours after completion of surgery. Hospital stay will be counted from the time the patient leaves the operating room to the time she leaves the hospital.

SECONDARY OUTCOMES:
Re-catheterization | Upto 4 weeks
  To demonstrate that immediate removal of catheter after minimally invasive sacrocolpopexy confers no increased risk of re-catheterization.
Urinary tract infection | upto 4 weeks
  To demonstrate that immediate removal of catheter after minimally invasive sacrocolpopexy decreases the occurrence of urinary tract infection.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad F Aslam, MD, Principal Investigator — St. John Hospital & Medical Center
Locations (3):
- United States (3):
  - St John Hospital & Medical Center, Detroit, Michigan
  - Oregon Health & Science University, Portland, Oregon
  - Legacy Good Samaritan Medical Center, Portland, Oregon

REFERENCES:
- [Derived] Ellahi A, Stewart F, Kidd EA, Griffiths R, Fernandez R, Omar MI. Strategies for the removal of short-term indwelling urethral catheters in adults. Cochrane Database Syst Rev. 2021 Jun 29;6(6):CD004011. doi: 10.1002/14651858.CD004011.pub4. PMID 34184246
- [Derived] Aslam MF, Bazzi AA, Hagglund KH, Osmundsen BC. When to Remove the Indwelling Catheter After Minimally Invasive Sacrocolpopexy? CARESS (CAtheter REmoval after Sacrocolpopexy Surgery). Female Pelvic Med Reconstr Surg. 2020 Feb;26(2):120-127. doi: 10.1097/SPV.0000000000000826. PMID 31990800